CLINICAL TRIAL: NCT04121130
Title: Shockwave Effectiveness in Myofascial Pain of the Upper Trapezius Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Garcia Cugat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REHA-2019-03
Record Dates: First submitted 2019-07-25; First posted 2019-10-09 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (F-ESWT Group) (Active Comparator): 3 F-ESWT sessions, 1 per week (0,10 mJ/mm2; 2000 impulses; 5 Hz) in the most painful tender and/or trigger points of the upper trapezius muscle.
  Interventions: Device: F-ESWT Group
- Group B (sham F-ESWT): (Placebo Comparator): 3 sham F-ESWT sessions, 1 per week (0,01 mJ/mm2; 2000 SW; 5 Hz) in the most painful tender and/or trigger points of the upper trapezius muscle.
  Interventions: Device: sham F-ESWT

INTERVENTIONS:
Device: F-ESWT Group — 3 F-ESWT sessions, 1 per week (0,10 mJ/mm2; 2000 impulses; 5 Hz) in the most painful tender and/or trigger points of the upper trapezius muscle.
  Arms: Group A (F-ESWT Group)
Device: sham F-ESWT — 3 sham F-ESWT sessions, 1 per week (0,01 mJ/mm2; 2000 SW; 5 Hz) in the most painful tender and/or trigger points of the upper trapezius muscle.
  Arms: Group B (sham F-ESWT):

SUMMARY:
Focused shockwaves are generated electrically, either within the applicator (electrohydraulic technique), or externally to it in the focal zone (electromagnetic or piezoelectric techniques), and then propagate to a designated focal point in order to treat it. Most research in shockwave therapy has focused on understanding the mechanism which results in the establishment of a mechano-sensitive feedback loop between the acoustic impulse and the stimulated cells, and involves specific transduction pathways and gene expression. Taking as valid the current physiopathological hypothesis of myofascial pain (MPS) and considering the mechanotransduction effect of ESWT in other diseases, it could be posited that ESWT in MPS may increase perfusion, promote angiogenesis and alter the pain signaling in ischaemic tissues caused by the influx of calcium. On the other hand, recent articles have demonstrated that free nerve endings degenerate after the application of ESWT, and that ESWT produces a transient dysfunction of nerve excitability at the neuromuscular junction, by bringing about the degeneration of AChR. Finally, following a pure mechanistic approach, shockwaves might be able to break-up the Actine-myosin links, as they are propagating perpendicularly to the sarcomere contractions.

Study Hypothesis: To obtain pain relief and improvement in functional and quality of life scales, by performing 3 ESWT sessions, 1 per week (0,10 mJ/mm2; 2000 impulses; 5 Hz) in the most painful tender and/or trigger points of the upper trapezius muscle.

Primary objective: To analyze the effectiveness of Focused Shockwave Treatment in myofascial pain of the upper trapezius muscle.

DETAILED DESCRIPTION:
This is a single blind randomized clinical trial that will be conducted in Quirónsalud Barcelona, Spain. The study will enroll 60 patients suffering of myofascial pain of the upper trapezius muscle over a 5-months period. The overall duration of the trial will be approximately 8 months. The trial will end when the last subject has the last visit, at 12 weeks (3 months).

This protocol calls for 7 visits to be performed over a 12-weeks period for each patient.

This study will enroll 60 patients suffering of myofascial pain of the upper trapezius muscle.

Treatment Assignment Procedures i. Randomization Procedures: The investigators will use block randomization, which is commonly used in the two treatment situations where the samples of the two treatments must be equal or equally equal. The process will involve recruiting participants in short blocks and ensuring that half of the participants within each block are assigned to "A" and the other half to "B". Within each block, however, the order of patients will be random. The patients will be considered blocks of four dimensions: 1. AABB, 2. ABAB, 3. ABBA, 4. BAAB, 5. BABA, 6. BBAA. The investigators will randomly select between these six different blocks for each group of four recruited participants. The random selection will be done using a list of random numbers generated using statistical software (Excel).

ii. Masking Procedures: The participants will be blinded to the type of ESWT treatment and the assessor, data managers, statistician and study monitors will be blinded to the allocation. All participants who receive ESWT treatment will be treated using the same device (Duolith® SD-1 STORZ Medical, Switzerland) regardless of what group patients are included in. The participants will not be able to predict the allocated group based on the appearance of the ESWT treatment. The blinding will be maintained until the data are locked. For blinding evaluation, allocation guessing will be assessed immediately after the final treatment. Practitioners and assessors will be instructed to treat the participants according to predefined standard operating procedures during the trial to maintain blinding.

Patients suffering of myofascial pain of the upper trapezius muscle, will be selected for this study, sign up for an informed consent form, informed about the details of the procedure and the potential risks before treatment and randomized into 2 treatment groups:

* Group A (F-ESWT group): 3 sessions, one per week, of focused extracorporeal shockwave treatment (2000 impulses at 0.10 mJ/mm2 per session).
* Group B (placebo group): 3 sessions, one per week, of sham focused extracorporeal shockwave treatment (2000 impulses at 0.01 mJ/mm2 per session).

All treatments will be performed by the senior authors. In all cases, a focused electromagnetic shockwave device will be used (Duolith® SD-1, STORZ Medical, Switzerland).

The procedure will be performed with the patient in sitting position, while the patient is lying in a pillow. The treatment area will be prepared with a coupling ultrasound gel to minimize the loss of shockwave energy at the interface between the tip of the applicator and the skin. No local anesthesia will be applied.

Post-treatment protocol All patients will receive a specific exercise protocol that includes home exercises and ergonomic indications to prevent an exacerbation of upper trapezius myofascial pain.

STUDY EVALUATIONS

Algometric Evaluation (PA): Pressure algometry [PA] is employed for quantification of tenderness in diagnosis of tender spots, trigger points, fibromyalgia and muscle spasm. The pressure pain threshold [PPT], i.e., the minimum pressure that induces pain or discomfort expresses the degree of sensitization affecting the nerve fibers by sensitizing substances. It offers the possibility to make a quantification of tenderness in myofascial and other musculoskeletal pain.

Visual Analogue Scale (VAS): The visual analogue scale (VAS) is considered to be one of the best methods available for the estimation of the intensity of pain. The VAS provides a continuous scale for magnitude estimation and consists of a straight line, the ends of which are defined in terms of the extreme limits of pain experience. Respondents mark the location on the 10-centimeter line corresponding to the amount of pain experienced. This gives the greatest freedom to choose pain's exact intensity. It also gives the maximum opportunity for each respondent to express a personal response style. VAS data of this type is recorded as the number of millimeters from the left of the line with the range 0-100.

Roles and Maudsley (RM): The RM scale is a subjective 4-point patient assessment of pain and limitations of activity.30 The RM score has been used extensively at centers throughout the world to assess outcome after SWT. On the scale, 1 point indicates an excellent result with the patient having no symptoms. Two points indicate a good result with the patient significantly improved from the pretreatment condition and satisfied with the result. Three points indicate a fair result with the patient somewhat improved from the pretreatment condition and partially satisfied with the treatment outcome. Four points indicate a poor outcome with symptoms identical or worse than the pretreatment condition and dissatisfaction with the treatment result.

EuroQol five dimensions questionnaire (EQ-5D-3L): The EQ-5D is a standardized measure of health status developed by the EuroQol Group to provide a simple, generic measure of health for clinical and economic appraisal. It is a simple questionnaire designed for completion by the person being treated.

EuroQol five dimensions VAS (EQ-5D-3L VAS): The EQ-5D VAS is a standardized measure of global health status, defined trough a scale from 0 (worst health status) from 100 (best health status).

Likert scale (1-6): Degree of recovery compared with baseline, measured on a 6-point Likert scale (completely recovered to much worse). Success rates will be calculated by dichotomizing responses. Subjects who will report themselves completely recovered or much improved will be counted as successes, and subjects who will report themselves somewhat improved, same, worse, or much worse will be counted as failures.

STATISTICAL CONSIDERATIONS

Efficacy variables Efficacy analyses will be performed on the sample group. Techniques of missing data handling, if applicable, will be described in the Statistical Analysis Plan.

Primary efficacy variable

1. Pain
2. Health status

Evaluation tools:

- Algometric evaluation (by pressure algometer)

Evaluation scales:

1. VAS
2. Roles and Maudsley
3. EQ-5D-5L INDEX VALUE
4. EQ VAS

Secondary efficacy variables

1. Agreement to the treatment

Evaluation scale: Likert scale

ETHICS/PROTECTION OF HUMAN SUBJECTS

1. Ethical Standard: This clinical study was designed and shall be conducted and reported in accordance with the International Conference for Harmonization (ICH) Harmonized Tripartite Guidelines for Good Clinical Practice, with applicable local regulations (including European Directive 2001/20/EC), and with the ethical principles laid down in the Declaration of Helsinki.
2. Independent Ethics Committee: The protocol, informed consent form, recruitment materials, and all subject materials will be submitted to an Independent Ethics Committee (IEC) in each center for review and approval. Approval of both the protocol and the consent form must be obtained before any subject is enrolled. The implementation of any change in the protocol will not be permitted until the principal investigator and the IEC have provided written approval of the change.
3. Informed Consent Process: Informed consent is a process that is initiated prior to the individual agreeing to participate in the study and continues throughout study participation. An extensive discussion of the risks and possible benefits of study participation will be held with the subjects. A consent form describing in detail the study procedures and risks will be given to the subject. Consent forms will be IEC-approved, and the subject is required to read and review the document or have the document read to him or her. The investigator or designee will explain the research study to the subject and answer any questions that may arise. The subject will sign the informed consent document prior to any study-related assessments or procedures. Subjects will be given the opportunity to discuss the study with their families and take all the time patients need prior to agreeing to participate. The patients may withdraw consent at any time throughout the course of the study. A copy of the signed informed consent document will be given to the subjects for their records. The rights and welfare of the subjects will be protected by emphasizing to them that the quality of their clinical care will not be adversely affected if the subjects decline to participate in this study. The consent process will be documented in the clinical records.
4. Subject Confidentiality: Subject confidentiality shall be guaranteed at all times by the investigators, study staff, and the sponsor and their delegates. The study protocol, documentation, data, and all other information generated will be strictly confidential. No information concerning the study or the data will be released to any unauthorized third party without prior written approval of the sponsor.

The study monitor or other authorized representatives of the sponsor may inspect all study documents and records required to be maintained by the investigator, including but not limited to the medical records of the study subjects. The clinical study site will permit access to such records.

DATA HANDLING AND RECORD KEEPING All study data are to be recorded on a database. All patient data shall be reported on the database in an anonymous fashion, the patient only being identified by the patient number.

The investigator will be responsible for the completeness, accuracy and timeliness of the data reported. All source documents should be completed in a neat, legible manner to ensure the accurate interpretation of data. The Investigator is required to verify the data transcribed onto the database.

The study monitors then have to check the database against the source documents for accuracy and validity as per the monitoring schedule, as applicable.

a. Data Management Responsibilities Data collection and accurate documentation are the responsibility of the study staff under the supervision of the investigator. All source documents and laboratory reports must be reviewed by Site staff and data entry staff, who will ensure that they are accurate and complete. Unanticipated problems and adverse events must be reviewed by the investigator or designee.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* No range of motion restriction
* Informed consent signed
* Diagnosis of myofascial pain of the upper trapezius muscle.
* Myofascial pain of the upper trapezius muscle non-responsive to physioterapic treatments

Exclusion Criteria:

* Age < 18 years
* Restricted range of motion
* Tumor in the area to be treated
* Wound in the area to be treated
* Coagulation disorders or anticoagulant therapy
* Local infection
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Algometric evaluation | 12 weeks
  Pressure algometry [PA] is employed for quantification of tenderness in diagnosis of tender spots, trigger points, fibromyalgia and muscle spasm.
VAS (Visual Analogue Scale) | 12 weeks
  The visual analogue scale (VAS) is considered to be one of the best methods available for the estimation of the intensity of pain.
Roles and Maudsley | 12 weeks
  The RM scale is a subjective 4-point patient assessment of pain and limitations of activity. The RM score has been used extensively at centers throughout the world to assess outcome after SWT.
EuroQol five dimensions questionnaire | 12 weeks
  The EQ-5D is a standardized measure of health status developed by the EuroQol Group to provide a simple, generic measure of health for clinical and economic appraisal.
EQ VAS | 12 weeks
  The EQ-5D VAS is a standardized measure of global health status.

SECONDARY OUTCOMES:
Likert scale | 12 weeks
  Degree of recovery compared with baseline, measured on a 6-point Likert scale (completely recovered to much worse). Success rates will be calculated by dichotomizing responses.

CONTACTS AND LOCATIONS:
Overall Officials: Montse García, Study Chair — Fundación García Cugat
Locations (1):
- Fundacion Garcia Cugat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No